CLINICAL TRIAL: NCT00577512
Title: 2006-32: Phase II Study of Rapidly Recycled High Dose DTPACE (HD-DTPACE) for Untreated or Previously Treated, High-Risk Multiple Myeloma (MM)
Brief Title: 2006-32 Phase II Study of Rapidly Recycled High Dose DTPACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-32
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2011-05-13 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HD DTPACE (Experimental): DTPACE
  Interventions: Drug: DTPACE

INTERVENTIONS:
Drug: DTPACE — * Dexamethasone 200 mg Intravenous Infusion "Piggy-Back" (IVPB) Days 1-7
  * Thalidomide 200 mg by mouth (PO) Days 1-7
  * Cisplatin 15mg/m2 Days 1-4 (modify for renal insufficiency)
  * Adriamycin 15 mg/m2 Days 1-4
  * Cyclophosphamide 600 mg/m2 Days 1-4
  * Etoposide 60 mg/m2 Days 1-4

SUMMARY:
This study is being done in an attempt to improve the remission rate and the survival time for subjects with high-risk myeloma. It is hoped that by giving higher doses of commonly used chemotherapy drugs and by giving courses closer together (before the myeloma comes back or gets worse), subjects in this study will have better outcomes.

DETAILED DESCRIPTION:
This study has the following goals:

* To find out how many subjects treated with high dose DTPACE (Dexamethasone, Thalidomide, CisPlatin, Adriamycin, Cyclophosphamide, and Etoposide. (HD DTPACE) on this protocol will have a complete response or near complete response that lasts for 6 months or longer.
* In subjects achieving a response, to find out how long the response will last.
* To learn more about the side effects of this treatment.

Up to 75 subjects, male or female, age 18 and older, regardless of race or ethnicity, will participate in this study at the University of Arkansas for Medical Sciences (UAMS) only.

The treatment in this study is divided into 3 parts

* High dose DTPACE and stem cell collection if you do not already have sufficient stem cells stored.
* High dose DTPACE and stem cell re-infusion.
* Velcade, Thalidomide, Dexamethasone (sometimes known as VTD) Maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma, treated or untreated, with the presence of one or more of the high risk features as defined below.

High risk by gene expression profiling at any time prior to enrollment:

1. PROLIFERATION signature, MMSET/FGFR3, c-MAF/MAF-B gene groups or
2. High risk score based on University of Arkansas Myeloma Institute for Research and Therapy (MIRT) 70 gene model.

   * Abnormal metaphase cytogenetics at any time prior to enrollment, or
   * Lactate Dehydrogenase (LDH) > 250 IU/L (upper limit normal) at any time prior to enrollment

     * Zubrod ≤ 2, unless due to symptoms of MM.
     * Patients must be < 75 years of age at the time of registration.
     * Patient must have signed an Institutional Review Board (IRB)-approved informed consent and understand the investigational nature of the study.
     * Negative serology for HIV.
     * Patients must not have a history of chronic obstructive or chronic restrictive pulmonary disease. Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, forced vital capacity (FVC), etc) and diffusion capacity (DLCO) > 50% of predicted. Patients unable to complete pulmonary function tests because of myeloma-related chest pain, must have a high resolution CT scan of the chest and must also have acceptable arterial blood gases defined as P02 greater than 70.
     * Patients with recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias are ineligible. Ejection fraction by echocardiogram (ECHO) or must be > 40% and must be performed within 60 days prior to registration, unless the patient has received chemotherapy within that period of time (dexamethasone and thalidomide excluded), in which case the left ventricular ejection fraction (LVEF) must be repeated.
     * No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years. Prior malignancy is acceptable provided there has been no evidence of disease within the three-year interval or if the malignancy is considered much less life threatening than the myeloma.
     * Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
     * Patients must be able to receive full doses of HD-DTPACE, in the opinion of the treating investigator, with the exception that patients with serum creatinine > 1.5 mg/dL will receive modified doses of cisplatin.

Exclusion Criteria:

* Fever or active infection requiring intravenous antibiotics within 72 hours from baseline.
* Liver function abnormalities with total bilirubin more than twice the upper limit of normal or aspartate amino transferase (AST)/alanine amino trasferase (ALT) more than three times the upper limit of normal.
* Severe renal dysfunction, defined as a creatinine > 3mg/dl or a creatinine clearance of <30ml/min.
* Platelet count < 30,000/mm3, or absolute neutrophil count (ANC) < 1,000/μl.
* Clinically significant hepatic dysfunction as noted by direct bilirubin or AST >3 times the upper normal limit or clinically significant concurrent hepatitis.
* New York Hospital Association (NYHA) Class III or Class IV heart failure.
* Poorly controlled hypertension, diabetes mellitus, or other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Prior adriamycin exposure > 450 mg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HD DTPACE: 1. High dose DTPACE (dexamethasone 200 mg days 1-7; thalidomide 200 mg days 1-4; cisplatin 15 mg/m2 days 1-4; adriamycin 15 mg/m2 days 1-4; cyclophosphamide 600 mg/m2 days 1-4; etoposide 60 mg/m2 days 1-4) and stem cell collection if you do not already have sufficient stem cells stored
  2. High dose DTPACE and stem cell re-infusion repeated every 18-21 days for 4 cycles
  3. Bortezomib (1.0 mg/m2 Day 1, 4, 8, 11), thalidomide (100 mg/m2 days 1-21), and dexamethasone (20 mg days 1-4 and 9-12) (VTD) Maintenance therapy
Period: Overall Study
Arm/Group | HD DTPACE
Started | 4
Completed | 0
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- HD DTPACE: 1. High dose DTPACE and stem cell collection if you do not already have sufficient stem cells stored
  2. High dose DTPACE and stem cell re-infusion
  3. VTD Maintenance therapy
Arm/Group | HD DTPACE
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Treated With (HD DTPACE Obtain a Complete Response or Near Complete Response That Lasts for 6 Months or Longer.
Description: Complete Response (CR) defined as all of the following for a minimum of 2 months: a) absence of urine and serum M-components by immunofixation; b) bone marrow should be adequately cellular (>20%); c) normal serum calcium; d) no new bone lesions or enlargement of existing lesions.
  Near Complete Response included all elements of CR except immunofixation studies remained positive.
Time Frame: 12 months
Measure: Number; unit: participant response
Arm/Group | HD DTPACE
Number analyzed (Participants) | 4
participant response | 0

ADVERSE EVENTS:
Arm/Group | HD DTPACE
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD DTPACE (N=4)
hypoxemia (General disorders) | 1 (1)
DVT (Blood and lymphatic system disorders) | 1 (4)
cellulitis (General disorders) | 1 (1)
pneumonia (General disorders) | 1 (1)
shortness of breath, cough, extreme weakness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes